CLINICAL TRIAL: NCT05749289
Title: Application of Al18F-octreotide PET/CT in Neuroendocrine Tumor
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NCC 3744
Record Dates: First submitted 2023-02-19; First posted 2023-03-01 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Neuroendocrine Tumor
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Al18F-NOTA-octreotide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Al18F-octreotide PET/CT (Experimental): Al18F-octreotide PET/CT will be performed on patients with suspected or clearly diagnosed Neuroendocrine Tumor. The patients were injected with Al18F-octreotide and underwent PET/CT scan 20~40min after the injection.
  Interventions: Drug: Al18F-octreotide

INTERVENTIONS:
Drug: Al18F-octreotide — Al18F-octreotide I was injected into the patients before the PET/CT scans
  Other Names: Al18F-NOTA-TATE

SUMMARY:
This is an open-label whole-body PET/CT study for investigating the value of Al18F-octreotide PET/CT in patients with Neuroendocrine Tumor

DETAILED DESCRIPTION:
Octreotide is an artificial replacement for the natural growth hormone inhibitor in humans. It is a small peptide hormone consisting of 14 amino acids and is widely distributed in neuroendocrine cells, with the highest density in the brain, peripheral neurons, endocrine pancreas and gastrointestinal tract. Under pathological conditions, some tumour cells show overexpression of growth inhibitory receptors, such as endocrine tumours of the pancreas, pituitary adenomas, pheochromocytomas, paragangliomas, carcinoid tumours, medullary thyroid carcinomas, small cell lung carcinomas and other neuroendocrine tumours. Therefore, the sensitivity and specificity of octreotide imaging is high.

This study will provide a visual, reproducible and non-invasive imaging method for the diagnosis of neuroendocrine tumours through Al18F-octreotide PCT/CT imaging, providing an intuitive and clear imaging basis for clinical diagnosis, differential diagnosis and treatment, contributing to the development of medicine and science in the field of positron imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected or clearly diagnosed Neuroendocrine Tumor
* signed written consent.
* Willing and able to cooperate with all projects in this study.

Exclusion Criteria:

* pregnancy;
* breastfeeding;
* any medical condition that in the opinion of the investigator may significantly interfere with study compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value | through study completion, an average of 1 year]
  Sensitivity and Specificity of Al18F-octreotide PET/CT for Neuroendocrine Tumor

CONTACTS AND LOCATIONS:
Overall Officials: Rong Zheng, M.D., Study Director — National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and PUMC
Locations (1):
- National Cancer Center/Cancer Hospital,Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Chao Yang, China

IPD SHARING:
Plan to Share IPD: No